CLINICAL TRIAL: NCT04453657
Title: Adapting and Delivering a Tele-Wellness Supported Digital Toolkit to Baltimore City's Approved Family Child Care Home Providers Caring for Children of Essential Workers: Promoting Health, Early Literacy, and Quality Parent Engagement Amid COVID-19: A Pilot Study
Brief Title: Tele-Wellness Supported App for Family Child Care Home Providers and Families to Promote Health, Family Engagement, and School Readiness Amid COVID-19
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00250864
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stress, Psychological; Child Behavior; Social Competence
Keywords: Family Child Care Home Providers; Parents; Young Children; Multi-component Self-Care; Tele-Wellness Service; Child care provider stress; Child care provider informational support; Behavior and Social functioning in Children; Educational learning games; Parent Engagement; Early Learning Intervention; Parenting; Social emotional learning games
MeSH Terms: conditions — Stress, Psychological; Child Behavior; Social Skills; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): There is only one arm in this study. All recruited and consented participants will fill out a pre-survey, engage with the digital toolkit for 15 weeks, then fill out a post-survey.
  Interventions: Device: FamilyChildCare (provisional name of app)

INTERVENTIONS:
Device: FamilyChildCare (provisional name of app) — Parents will provide their child(ren) access to a smartphone, tablet, or computer for approximately 30 minutes, three times per week for 15 weeks with a total dosage of instruction of about 22.5 hours. Parents and providers will receive self-care, parenting, and parent engagement tips and resources through push notifications twice a day. Additionally, daily reminders will be sent to parents through push notification to give their child(ren) access to the learning games. After 15 weeks of app engagement, the providers and parents will be contacted by the PI to notify them of the 15 week time mark and provide the information for post-surveys via Qualtrics.

SUMMARY:
The investigators aim to deliver a tele-wellness supported app to Baltimore City's Family Child Care Home (FCCH) providers who are caring for children of Essential Personnel. Once a pre-survey is conducted, login information will be assigned to 30 Family Child Care Home providers and parents the FCCH serve. Providers and Parents will receive self-care and parenting/parent engagement support through the app and through a tele-wellness service, Ask a Nurse, provided by community health nurses at the Johns Hopkins School of Nursing. Children will have access to gamified learning materials in early literacy, math, social-emotional learning, and nutrition.

DETAILED DESCRIPTION:
The investigators will adapt and deliver a tele-wellness supported digital toolkit via an app for Baltimore City's Family Child Care Home (FCCH) providers and the families the FCCH serve. Through this digital toolkit, the investigators aim to provide related self-care support, parent/parent engagement support for both Family Child Care Home providers and parents, and provide access to early literacy, math, social-emotional learning, and nutrition games for children (3-6 years old). Additionally, Family Child Care Home providers and parents will have access to a hotline and email to the Ask a Nurse program-a tele-wellness program run by community registered nurses at Johns Hopkins School of Nursing. Through Ask a Nurse, providers and parents will be able to receive wellness counseling from licensed registered nurses and care coordination to address specific social needs. The tele-wellness service is NOT intended to directly address health issues, diagnose, or prescribe. In summary, Family Child Care Home providers will have access to self-care and parent engagement resources and parents will have access to self-care and parenting resources in addition to the games for the child(ren).

The first phase of this study is to tailor an existing app, Escribo Play that already has gamified early literacy and math tools, and expand its scope by including self-care and parenting/parent engagement support for Family Child Care Home Providers and the parents the FCCH serve. Additionally, the investigators are creating gamified social-emotional learning and nutrition games for the children.

The second phase is a pre-post test where the investigator will recruit FCCH providers enrolled in the Essential Personnel Child Care or School-Aged program and the parents the FCCH serve to fill out health surveys before and 15 weeks post engagement with the app.

The investigators hypothesize that engagement with the digital toolkit will improve provider and parental perceived level of stress, informational support, access to learning games, as well as social, emotional, and behavioral functioning in children.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Family Child Care Home Providers operating in Baltimore City who are approved or was once approved to remain open during COVID-19 through the Essential Personnel Child Care or School-Aged Program.
* Parents or legal adult guardians of young children (3-6 years old) who have utilized or continue to utilize the services of Family Child Care Home providers enrolled in the study.
* All participants must have access to a smartphone, tablet, or computer.

Exclusion Criteria:

* Licensed Family Child Care Home Providers not enrolled or was never enrolled in the Essential Personnel Child Care or School-Aged Program
* Parents of young children (3-6 years old) who have not utilized the services of Licensed Family Child Care Home Providers in the Essential Personnel Child Care or School-Aged Program
* FCCH providers not operating in Baltimore City
* FCCH providers who do not have at least 1 parent consenting to participate in the study.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Level of Stress as assessed by the Perceived Stress Scale | At pre and post surveys lasting 30-45 minutes each, up to 15 weeks apart
  Family Child Care Home Providers & Parents: Perceived Stress Scale (PSS)-10 is a 10-item tool widely used to measure the degree to which circumstances in one's life are deemed as stressful in the general population. The PSS was designed for use in community samples with at least a junior high school education. The items are easy to understand, and the response alternatives are simple to grasp. Six items of the PSS-10 are negatively phrased (item 1, 2, 3, 6, 9, 10; negative perception subscale, while the remaining four (item 4, 5, 7 and 8; positive perception subscale) are positively phrased items and require reverse coding. Total PSS-10 score will be calculated by summing scores. A total score ranges 0-40 where a higher score indicates higher perceived stress.
Change in Perceived Level of Informational Support as assessed by the PROMIS Informational Support Short Form | At pre and post surveys lasting 30-45 minutes each, up to 15 weeks apart
  Family Child Care Home Providers & Parents: Patient-Reported Outcomes Measurement Information System (PROMIS) Informational Support Short Form 8a assesses the perceived availability of helpful information or advice. It is an 8-item tool and each item has 5 response options ranging in values from one to five-1=Never 2=Rarely 3=Sometimes 4=Usually 5=Always with a range of 8-40. Total raw scores, sum of values to responses, will be calculated. A Score conversion table found in the Appendix of the tool will be used to translate the total raw score or pro-rated score into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Change in Awareness of the Maryland Early Childhood Family Engagement Framework and Toolkit as assessed by a survey question | At pre and post surveys lasting 30-45 minutes each, up to 15 weeks apart
  Family Child Care Home providers will be asked in the pre/post-surveys whether they are aware of the existence of the Maryland Early Childhood Family Engagement Framework and Toolkit- a 91-page document developed by the Maryland State Department of Education to guide child care providers in best practices for family engagement. Family Child Care Home providers will respond either
  i. Yes, I am aware of it but have not read it ii. Yes, I am aware of it and have read the report iii. No, I am not aware of it
Change in Social, Emotional, and Behavior Functioning in Children as assessed by the Social Competence and Behavior Evaluation for Children | At pre and post surveys lasting 30-45 minutes each, up to 15 weeks apart
  The social, emotional, and behavioral functioning in children will be assessed by parents responding to items on the Social Competence and Behavior Evaluation for Children: The Short Form (SCBE)-30. It is a 30 item tool with a 6 point response option- Never (1), Sometimes (2 or 3), Often (4 or 5), or Always (6). The SCBE-30 has three subscales (10 items each): Anger-Aggression (cronbach's α = 0.93 in the current sample), Anxiety-Withdrawal (cronbach's α = 0.87), and Social Competence (cronbach's α = 0.89). The SCBE-30 was developed for children from ages three to six and has been shown to have high interrater and test-retest reliability and internal consistency. Sums of each subscale will be calculated.

SECONDARY OUTCOMES:
Change in Quality of the Parent-Child Care Relationship as assessed by the Supportive Parent-Caregiver Relationship Subscale | At pre and post surveys lasting 30-45 minutes each, up to 15 weeks apart
  Family Child Care Home Provider and Parents: The Supportive Parent-Caregiver Relationship Sub-scale from Scales Measuring Aspects of Child-Care Quality Supportive Parent-Caregiver Relationship assess the perceived quality of the Parent-Child Care Relationship. The provider report contains 6 items with a 5 point response scale-1=Never, 2=Rarely, 3=Sometimes, 4=Often, or 5=Always. The scale will be adapted to ask about the general relationship to all parents, not any specific parent. The parent report contains 6 items with a 5 point response scale-1=Never, 2=Rarely, 3=Sometimes, 4=Often, or 5=Always. The mean score & alpha will be reported. Reported Mean=26.9, SD=3.4, Alpha=.84)

CONTACTS AND LOCATIONS:
Overall Officials: Lucine Francis, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No